CLINICAL TRIAL: NCT05684380
Title: National, Multicenter, Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of MAZ-101 in the Treatment of Persistent Allergic Rhinitis (PER)
Brief Title: Efficacy and Safety of MAZ-101 in the Treatment of Persistent Allergic Rhinitis (PER)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0422 - AZALEIA
Record Dates: First submitted 2022-12-16; First posted 2023-01-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAZ-101 (Experimental): One applications in each nostril, twice a day.
  Interventions: Drug: MAZ-101association
- DYMISTA® (Active Comparator): One applications in each nostril, twice a day.
  Interventions: Drug: DYMISTA®

INTERVENTIONS:
Drug: MAZ-101association — Experimental drug
  Arms: MAZ-101
Drug: DYMISTA® — Active comparator
  Arms: DYMISTA®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MAZ-101 in the treatment of moderate-severe persistent allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes, with age greater than or equal to 12 years;
* Clinical diagnosis of moderate-severe persistent for at least 1 year;
* Screening Visit: A 12-hour reflective TNSS ≥ 8 out of a possible 12 and a congestion score of 2 or 3;
* Randomization Visit: A 12-hour reflective TNSS (AM or PM) ≥ 8 on 3 separate symptoms assessments during the Lead-in Period; an AM or PM 12-hour reflective nasal congestion score of 2 or 3 must have been recorded on 3 separate symptom assessments;
* Present skin sensitization test to at least one aeroallergen.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Other clinical forms of rhinitis;
* Subjects receiving immunotherapy;
* Presence of nasal polyposis;
* Patients with severe arterial hypertension, severe coronary diseases, cardiac arrhythmias, glaucoma, ocular herpes simplex, cataracts, hyperthyroidism;
* Asthma sufferers; respiratory tract infections and lung disease, including chronic obstructive pulmonary disease (COPD);
* Presence of grade II or III septal deviation and/or presence of nasal polyps or other conditions that determine nasal obstruction;
* Concomitant chronic or intermittent use of decongestants and/or antihistamines and/or inhaled, oral, intramuscular, intravenous or potent topical corticosteroids;
* Participants using monoamine oxidase inhibitors (MAOIs);
* Participants with known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* History of alcohol abuse or illicit drug use;
* Pregnancy or risk of pregnancy and lactating patients;

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in AM+PM rTNSS (reflective total nasal symptoms score). | 28 days.
  Change from baseline in 12-hour reflective total nasal symptom score (rTNSS) consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary for the entire 28 day study period. The measurement scale is 0 to 24 so that the higher the number the worse the symptom.

SECONDARY OUTCOMES:
Change from baseline in AM+PM rTOSS (reflective total ocular symptom score). | 28 days.
  Change from baseline in 12-hour reflective total ocular symptom score (rTOSS) consisting of itching/burning, tearing/watering, and redness scored twice daily (AM and PM) in diary for the entire 28 day study period. The measurement scale is 0 to 18 so that the higher the number the worse the symptom.
Change from baseline in AM + PM: rTNSS (reflective total nasal symptoms score) plus rTOSS (reflective total ocular symptom score). | 28 days.
  Change from baseline in 12-hour rTNSS plus rTOSS consisting of nasal congestion,runny nose, itchy nose and sneezing that represents rTNSS and itching/burning, tearing/watering, and redness that represents rTOSS scored twice daily (AM and PM) in diary for the entire 28 day study period. The measurement scale is 0 to 24 of rTNSS plus 0 to 18 of rTOSS. Then, the (rTNSS plus rTOSS ) measurement scale is 0 to 42 so that the higher the number the worse the symptom.
Change from baseline in reflective individual nasal symptom scores. | 28 days.
  Change from baseline in the 12-hour reflective individual nasal symptom scores consisting of nasal congestion,runny nose, itchy nose, sneezing scored twice daily (AM and PM) in diary for the entire 28 day study period. The measurement scale is 0 to 3 in each symptom so that the higher the number the worse the symptom.
Change from baseline in reflective individual ocular symptom scores. | 28 days.
  Change from baseline in the 12-hour reflective individual ocular symptom scores consisting of itching/burning, tearing/watering, and redness scored twice daily (AM and PM) in diary for the entire 28 day study period. The measurement scale is 0 to 3 in each symptom so that the higher the number the worse the symptom.
Change from baseline in the Rhinoconjunctivitis Quality of Life Questionnaire for adults (RQLQ) or Rhinoconjunctivitis Quality of Life Questionnaire for adolescents (AdolRQLQ). | 28 days.
  Change compared to baseline in the general score of the Adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) or adolescent (AdoRQLQ) after 28 days os treatment. The RQLQ has 28 questions and the AdolRQLQ has 25 questions. Participants will respond to each question on a 7-point scale (0 = not at all impaired to 6 = severely impaired) according to how bothered the participants were by their rhinoconjunctivitis during the past week.
Number of days without nasal symptoms | 28 days.
  Number of days without nasal symptoms (rTNSS = 0) for the entire 28-day study period.

IPD SHARING:
Plan to Share IPD: No